CLINICAL TRIAL: NCT04699162
Title: Efficacy of Intermediate and High Intensity Regimens in Patients With Relapsed Acute Lymphoblastic Leukemia. Experience of Two Centers in Mexico City
Brief Title: Efficacy of Intermediate and High Intensity Regimens in Patients With Relapsed Acute Lymphoblastic Leukemia
Acronym: HGMHRAEI/ALL
Status: Completed | Type: Observational
Sponsor: Christian Omar Ramos-Peñafiel, MD, PhD (Other Government)
Responsible Party: Sponsor-Investigator, Christian Omar Ramos-Peñafiel, MD, PhD, Head of the hematology hospitalization area, Hospital General de Mexico
Organization: Hospital General de Mexico (Other Government)
Other Study IDs: DECS/JPO-CT-397-2020
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Survival; Leukemia; Relapse; Retrospective study
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to describe the survival and relapses of patients with diagnosis of acute lymphoblastic leukemia at two tertiary level hospitals in the metropolitan area of the valley of Mexico

DETAILED DESCRIPTION:
Retrospective, observational study in patients with diagnosis of acute lymphoblastic leukemia, according to the criteria of the World Health Organization, from July, 2016, to October, 2020. The patients were cared for in the hematology department of the Hospital General de Mexico and in the hematology department of the Hospital Regional de Alta Especialidad Ixtapaluca. Relapse was considered in those cases with more than 5% of blasts in bone marrow and as relapse to the central nervous system with the presence of blasts in cerebrospinal fluid.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of acute lymphoblastic leukemia according to the criteria of the World Health Organization.

Exclusion Criteria:

* Age less than 15 years
* Age over 60 years

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with first diagnosis of acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 4-years
Progression free survival | 4-years
Number of relapses | 4-years
  Cases with more than 5 percent of blasts in bone marrow and as relapse to the central nervous system with the presence of blasts in cerebrospinal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Christian O Ramos-Peñafiel, MD, Ph.D, Principal Investigator — Hospital General de México Dr. Eduardo Liceaga
Locations (2):
- Mexico (2):
  - Hospital Regional de Alta Especialidad de Ixtapaluca, Ixtapaluca, State of Mexico
  - Hospital General de México "Dr. Eduardo Liceaga", Mexico City